CLINICAL TRIAL: NCT05671406
Title: A Sensor-controlled Digital Game-based Approach to Improve Self-care Behaviors Among Adults Diagnosed With Hypertension in a Native American Community
Brief Title: RCT of Sensor-controlled Digital Game for Hypertension Self-care in a Native American Community
Acronym: N-SCDG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Kavita Radhakrishnan, Principal Investigator, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: R01HL162598 (NIH); STUDY00002092 (Other: UT Austin IRB); R01HL162598 (NIH)
Record Dates: First submitted 2023-01-02; First posted 2023-01-04 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Hypertension
Keywords: hypertension; self-care; digital game; Native American
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensor-controlled digital game (Experimental): The intervention group will receive a sensor-controlled digital game (SCDG) app and physical activity tracker.
  Interventions: Behavioral: Sensor-controlled digital game
- Sensor-only (Active Comparator): The control group will receive only the physical activity tracker.
  Interventions: Behavioral: Sensor only

INTERVENTIONS:
Behavioral: Sensor-controlled digital game — The SCDG will involve a narrative, the goal of which is to help an avatar in the game avoid hospitalization by using game points, earned via the participant's real-time behaviors, in game tasks that help maintain the avatar's optimal Hypertension health status. Real-time behaviors of weight-monitoring and physical activity will be tracked by an off-the-shelf sensors and app (Withings). The data from the Withings sensors will then be routed to our SCDG app.
  The digital game paired with sensors will enable objective tracking of real-time behaviors such as physical activity, and weight monitoring, and provide personalized, contextually relevant feedback to motivate engagement in and generate habit formation of heart failure related self-management behaviors.
  Other Names: SCDG
  Arms: Sensor-controlled digital game
Behavioral: Sensor only — Real-time behaviors of physical activity will be tracked by an off-the-shelf sensor and app (Withings). This group will also be provided with standardized evidence-based Hypertension educational material. However, the data from the Withings sensor will not be routed to the SCDG.
  Arms: Sensor-only

SUMMARY:
This study evaluates a sensor-controlled digital game (SCDG) to motivate self-management behaviors of physical activity in Native American adults with hypertension (HTN). Half of the participants will receive the SCDG app and physical activity sensors and the other half will receive only the physical activity sensors.

Native American participants with hypertension (HTN) in the sensor controlled digital game intervention group will show increased PA behaviors; improved HTN knowledge, self-care behaviors, self-efficacy, motivation, and quality of life (QoL); and larger reduction in systolic and diastolic blood pressure and cardiac hospitalizations at baseline,3 months, and 6 months as compared to participants in the sensor-only control group.

DETAILED DESCRIPTION:
Cardiovascular disease is the leading cause of death among Native Americans (NAs). Hypertension (HTN) strongly elevates the morbidity and mortality risks related to cardiovascular disease. Lifestyle modifications promoted by U.S. HTN guidelines includes modifiable self-care behaviors such as regular physical activity which is associated with lower blood pressure, reduced cardiovascular risk, and beneficial cardiac structural remodeling. Therefore, motivating physical activity behaviors would be key to cardiovascular health promotion efforts among a Native American community.

One promising approach is the use of sensor-controlled digital games (SCDGs), which offer affordable, portable, and scalable tools to facilitate engagement in HTN self-care behaviors while being enjoyable and easy to use. The SCDG intervention integrates HTN participants' behavioral data from an activity tracker sensor to activate game progress, rewards, and feedback. The primary goal of this study is to test a culturally adapted SCDG intervention (N-SCDG) for improving daily physical activity self-care behaviors among Lumbee tribal adults with HTN and examine approaches for sustaining the impact of the N-SCDG at the community level.

The investigators will compare the N-SCDG intervention versus a sensor-only control for the primary outcome of engagement in the HTN selfcare behavior of physical activity and the secondary outcomes of HTN self-care knowledge, self-care behaviors, self-efficacy, systolic and diastolic blood pressure, cardiac hospitalization, and quality of life at baseline, 3 months, and 6 months. The investigators will randomize 220 participants to either the N-SCDG intervention group, in which participants will receive sensors that track physical activity and will play the N-SCDG on a mobile smart phone, or a control group that will receive sensors, an app that tracks physical activity, and standardized written HTN educational materials.

ELIGIBILITY:
Inclusion Criteria:

* Adults in a Native American tribal community in southeastern U.S.
* Age 18 years or older
* Systolic BP ≥140mm Hg and/or diastolic BP ≥90mm Hg on 2 separate measurements or who are on antihypertensive medication will be included.
* Pass a mini-cognitive screen
* Able to independently walk without using a walker or requiring human assistance (ambulation/locomotion item on the Outcome and Assessment Information).

Exclusion Criteria:

* Severe visual (e.g., legal blindness) or tactile (e.g., severe arthritis) impairments that adversely prevent use of a smart phone or sensor devices;
* Chronic kidney disease stage 4-5,
* Diagnosis of end stage or terminal illness (e.g., cancer or heart failure)
* Prior heart transplantation or implantation of a durable mechanical circulatory support device (e.g., left ventricular assist devise) due to unique self-care needs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Mean of Daily Steps on Physical Activity Sensor Logs at 3 months | 3 months
  This outcome measure will be measured by calculating the average daily steps at end of 3 months. These measures will be collected from sensor logs within the apps for both IG and CG.
Mean of Daily Steps on Physical Activity Sensor Logs at 6 months | 6 months
  This outcome measure will be measured by calculating the average daily steps at end of 6 months. These measures will be collected from sensor logs within the apps for both IG and CG.

SECONDARY OUTCOMES:
Change from baseline in Mean Systolic Blood Pressure as measured by a FDA approved digital sphygmomanometer at 3 months. | Baseline, 3 months
  Systolic blood Pressure (SBP) of participants will be measured at baseline using a FDA approved digital sphygmomanometer (A&D UA-767). The A&D UA-767 is a fully automated device based on the oscillometric method and has been validated against a mercury sphygmomanometer. Participants will be instructed to refrain from using tobacco products, alcohol, or caffeine for 30 minutes before measurement. Participants will sit quietly, resting the left arm on a flat surface (at the heart's level) for at least 5 minutes before the first measurement. Three measurements will be taken at 1-minute intervals; the second and third readings recorded in mmHg will be averaged to obtain the mean SBP.
Change from baseline in Mean Systolic Blood Pressure as measured by a FDA approved digital sphygmomanometer at 6 months. | Baseline, 6 months
  Systolic blood Pressure (SBP) of participants will be measured at baseline using a FDA approved digital sphygmomanometer (A&D UA-767). The A&D UA-767 is a fully automated device based on the oscillometric method and has been validated against a mercury sphygmomanometer. Participants will be instructed to refrain from using tobacco products, alcohol, or caffeine for 30 minutes before measurement. Participants will sit quietly, resting the left arm on a flat surface (at the heart's level) for at least 5 minutes before the first measurement. Three measurements will be taken at 1-minute intervals; the second and third readings recorded in mmHg will be averaged to obtain the mean SBP.
Change from baseline in Mean Diastolic Blood Pressure as measured by a FDA approved digital sphygmomanometer at 3 months. | Baseline, 3 months
  Diastolic blood Pressure (DBP) of participants will be measured at baseline using a FDA approved digital sphygmomanometer (A&D UA-767). The A&D UA-767 is a fully automated device based on the oscillometric method and has been validated against a mercury sphygmomanometer. Participants will be instructed to refrain from using tobacco products, alcohol, or caffeine for 30 minutes before measurement. Participants will sit quietly, resting the left arm on a flat surface (at the heart's level) for at least 5 minutes before the first measurement. Three measurements will be taken at 1-minute intervals; the second and third readings recorded in mmHg will be averaged to obtain the mean DBP.
Change from baseline in Mean Diastolic Blood Pressure as measured by a FDA approved digital sphygmomanometer at 6 months. | Baseline, 6 months
  Diastolic blood Pressure (DBP) of participants will be measured at baseline using a FDA approved digital sphygmomanometer (A&D UA-767). The A&D UA-767 is a fully automated device based on the oscillometric method and has been validated against a mercury sphygmomanometer. Participants will be instructed to refrain from using tobacco products, alcohol, or caffeine for 30 minutes before measurement. Participants will sit quietly, resting the left arm on a flat surface (at the heart's level) for at least 5 minutes before the first measurement. Three measurements will be taken at 1-minute intervals; the second and third readings recorded in mmHg will be averaged to obtain the mean DBP.
Change from baseline in mean Blood Pressure Control at 3 months | Baseline, 3 months
  Blood Pressure will be measured as described above for Systolic and Diastolic blood pressure. Blood Pressure Control will be defined as yes if mean SBP < 140 mmHG and mean DBP < 90 mmHG.
Change from baseline in mean Blood Pressure Control at 6 months | Baseline, 6 months
  Blood Pressure will be measured as described above for Systolic and Diastolic blood pressure. Blood Pressure Control will be defined as yes if mean SBP < 140 mmHG and mean DBP < 90 mmHG.
Change From Baseline in Hypertension Knowledge as measured by the Hypertension Knowledge-Level Scale (HK-LS) at 3 months | Baseline, 3 months
  Knowledge will be measured by the Hypertension Knowledge-Level Scale (HK-LS). The scale has 22 items with six sub-dimensions of definition, medical treatment, drug compliance, lifestyle, diet, and complications, respectively. Each correct answer is worth 1 point. The maximum scale score is 22, being scored only when the respondent provides the right answer. Higher scores indicate higher knowledge.
Change From Baseline in Hypertension Knowledge as measured by the Hypertension Knowledge-Level Scale (HK-LS) at 6 months | Baseline, 6 months
  Knowledge will be measured by the Hypertension Knowledge-Level Scale (HK-LS). The scale has 22 items with six sub-dimensions of definition, medical treatment, drug compliance, lifestyle, diet, and complications, respectively. Each correct answer is worth 1 point. The maximum scale score is 22, being scored only when the respondent provides the right answer. Higher scores indicate higher knowledge.
Change From Baseline in Hypertension self-efficacy as measured by the hypertension self-efficacy subscale of the High Blood Pressure Hypertension Self-Care Profile at 3 months | Baseline, 3 months
  The hypertension self-efficacy subscale of the High Blood Pressure Hypertension Self-Care Profile has 20 items. Items in this subscale include a 4-point scale format asking how confident are individuals in performing certain behaviors necessary to manage HTN (e.g., physical activity, nutrition). Responses were rated from 1 (not relevant) to 4 (very relevant). Scores are summed with higher scores indicating higher self-efficacy in managing HTN. Scores can range from 20 to 80.
Change From Baseline in Hypertension self-efficacy as measured by the hypertension self-efficacy subscale of the High Blood Pressure Hypertension Self-Care Profile at 6 months | Baseline, 6 months
  The hypertension self-efficacy subscale of the High Blood Pressure Hypertension Self-Care Profile has 20 items. Items in this subscale include a 4-point scale format asking how confident are individuals in performing certain behaviors necessary to manage HTN (e.g., physical activity, nutrition). Responses were rated from 1 (not relevant) to 4 (very relevant). Scores are summed with higher scores indicating higher self-efficacy in managing HTN. Scores can range from 20 to 80.
Change From Baseline in Hypertension self-care behaviors as measured by the hypertension behavior subscale of the High Blood Pressure Hypertension Self-Care Profile (HBP-SCP) at 3 months | Baseline, 3 months
  The hypertension behavior subscale of the High Blood Pressure Hypertension Self-Care Profile (HBP-SCP) has 20 items. Items in this subscale include a 4-point scale format asking how often individuals performed certain behaviors necessary to manage HTN (e.g., physical activity, nutrition). Responses were rated from 1 (not relevant) to 4 (very relevant). Scores were summed with higher scores indicating more positive self-care behaviors in managing hypertension. Scores can range from 20 to 80.
Change From Baseline in Hypertension self-care behaviors as measured by the hypertension behavior subscale of the High Blood Pressure Hypertension Self-Care Profile (HBP-SCP) at 6 months | Baseline, 6 months
  The hypertension behavior subscale of the High Blood Pressure Hypertension Self-Care Profile (HBP-SCP) has 20 items. Items in this subscale include a 4-point scale format asking how often individuals performed certain behaviors necessary to manage HTN (e.g., physical activity, nutrition). Responses were rated from 1 (not relevant) to 4 (very relevant). Scores were summed with higher scores indicating more positive self-care behaviors in managing hypertension. Scores can range from 20 to 80.
Change from Baseline in Quality of Life as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Global-10 at 3 months | Baseline, 3 months
  The PROMIS Global-10 is a 10-item questionnaire that assesses the general quality of life (QOL) divided into two domains-physical and mental health. Each domain's scores are derived using T-score normal population distribution mean ± standard deviation (SD) of 50 ± 10, where higher scores indicate better health.
Change from Baseline in Quality of Life as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Global-10 at 6 months | Baseline, 6 months
  The PROMIS Global-10 is a 10-item questionnaire that assesses the general quality of life (QOL) divided into two domains-physical and mental health. Each domain's scores are derived using T-score normal population distribution mean ± standard deviation (SD) of 50 ± 10, where higher scores indicate better health.
Number of Cardiac Hospitalizations in the past month at 3 months | Baseline, 3 months
  This measure will be obtained through participant self-report through periodic online surveys and will be confirmed by hospital discharge summary provided by the participant.
Number of Cardiac Hospitalizations in the past month at 6 months | Baseline, 6 months
  This measure will be obtained through participant self-report through periodic online surveys and will be confirmed by hospital discharge summary provided by the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Kavita Radhakrishnan, Phd, Principal Investigator — The University of Texas Austin
Locations (1):
- University of North Carolina Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
The investigators will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. After review of the purpose of the data request to make sure it is consistent with the original project goals and verification that the request meets IRB approval, de-identified data may be shared with researchers as soon as possible but no later than within one year from the completion of the funded project period for the parent award or upon acceptance of the data for publication, whichever is earlier.

REFERENCES:
- [Derived] Radhakrishnan K, Im CR, Brooks JL, Fallon GC, Rangel A, Julien C, O'Hair M, Liang H, Lowe J. Sensor-controlled digital game for Native American adults in the Lumbee Tribe with hypertension self-management: study protocol for a randomized controlled trial. Trials. 2025 Sep 1;26(1):329. doi: 10.1186/s13063-025-09026-y. PMID 40890750